CLINICAL TRIAL: NCT02297828
Title: Effect of Boussignac Continuous Positive Airway Pressure Ventilation on PaO2 and PaO2/FiO2 Ratio Immediately After Extubation in Morbidly Obese Patients Undergoing Bariatric Surgery: a Randomized Controlled Trial
Brief Title: Effect of Boussignac CPAP Ventilation on PaO2 and PaO2/FiO2 Ratio in Morbidly Obese Patients Undergoing Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Joana Alexandra Carvalho Guimarães, MD, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 278/13
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Boussignac CPAP (Experimental): Boussignac CPAP with a 50% FiO2 (adjusted in a piece adapted to the system) and a pressure of 5cmH2O (measured with a manometer) is applied immediately after extubation and mantained for two hours after extubation in the post anesthesia care unit (PACU).
  Arterial blood samples to measure PaO2 and PaO2/FiO2 ratio are collected before surgery and at 1, 2 and 24 hours after extubation. Spirometry is performed at the same intervals measuring FEV1 and FVC.
  Interventions: Device: Boussignac CPAP
- Ventury face mask (Active Comparator): Venturi mask with a 50% FiO2 is used immediately after extubation and mantained for two hours in the post anesthesia care unit (PACU).
  Arterial blood samples to measure PaO2 and PaO2/FiO2 ratio are collected before surgery and at 1, 2 and 24 hours after extubation. Spirometry is performed at the same intervals measuring FEV1 and FVC.
  Interventions: Device: Venturi face mask

INTERVENTIONS:
Device: Boussignac CPAP — Boussignac CPAP with a 50% FiO2 (adjusted in a piece adapted to the system) and a pressure of 5cmH2O (measured with a manometer) is applied immediately after extubation and mantained for two hours after extubation in the post anesthesia care unit (PACU).
  Arms: Boussignac CPAP
Device: Venturi face mask — Venturi mask with a 50% FiO2 is used immediately after extubation and mantained for two hours in the post anesthesia care unit (PACU).
  Arms: Ventury face mask

SUMMARY:
The purpose of this study is to determine if the application of Boussignac continuous positive airway pressure (CPAP) immediately after extubation improves PaO2 and PaO2/FiO2 ratio in morbidly obese patients undergoing gastric bypass surgery .

DETAILED DESCRIPTION:
Background: In 2010, the prevalence of obesity in individuals above 15 years old in Portugal was 15.5% for males and 17.7% for females. .In this country bariatric surgery has increased significantly playing an important role in the treatment of individuals with BMI ≥ 40 kg/m2 or less than 35 kg/m2 in the presence of comorbidities.

Morbid obesity has a negative impact in the respiratory physiology and is associated with a decreased compliance of the lung and chest wall, increased airway resistance, decreased respiratory muscle strength, increased work of breathing, worsening of ventilation / perfusion ratio and postoperative hypoxemia. General anesthesia and surgery in these patients will maximize these physiologic alterations.

Ahmad et al. (2008) found that morbid obesity per se, regardless of the presence of obstructive sleep apnea was associated with increased risk of desaturation in the first 24h of the postoperative period.

Gaszynski et al. (2007) found that the use of Boussignac CPAP in the postoperative period of patients undergoing bariatric surgery improved oxygenation. However, it was used capillary blood gas analysis not arterial blood and the FiO2 was different between groups.

More recently, in 2011, Wong et al. investigated the effect of Boussignac CPAP versus Venturi mask in the first one hour after bariatric surgery, measuring the PaO2 / FiO2 ratio at 1 hour and 2 hours of the postoperative period. The group maintained with CPAP showed better results. There were no differences between the two groups for FEV1 and FVC. The study does not reveal, however, the analgesic protocol used postoperatively or the patient's position during the spirometric measurements. These variables could be possible confounders. The PaO2 absolute value was not evaluated because of the different FiO2 between patients.

Objectives: We aim to assess the impact of the application of Boussignac CPAP ventilation immediately after extubation for improving PaO2 and PaO2/FiO2 ratio in morbidly obese patients submitted to gastric bypass surgery. As a secondary objective we intend to evaluate if there are differences in spirometry parameters.

Methods: A randomized controlled study on 24 patients undergoing gastric bypass surgery. Control group receives a Ventury mask immediately after extubation and the intervention group gets the Boussignac CPAP immediately after extubation. Both groups have the same anesthetic protocol during the intraoperative period and receive a 50% FiO2 after extubation. Venturi mask and Boussignac CPAP are maintained for two hours. A blood sample is collected from radial artery to measure PaO2 and calculate PaO2/FiO2 ratio before surgery and at 1, 2 and 24 hours after extubation in both groups. Evaluation of forced expiraroty volume in 1 second (FEV1) and forced vital capacity (FVC) with a portable spirometer is also performed at the same intervals. Patients are monitored for oxygen saturation, arterial pressure and cardiac rhythm while using the devices. Tolerance to the device, analgesic requirements and sedation level are also monitored and registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 65 years of age
* Morbidly obese with a body mass index > 35 kg/m2
* Laparoscopic gastric bypass

Exclusion Criteria:

* Patient refusal
* American Society of Anesthesiologists' (ASA) class IV
* Lung parenchyma disease
* Chronic Obstructive Pulmonary Disease
* Moderate to severe asthma
* Pre-existing cardiac failure (above class II in the New York Heart Association (NYHA) classification)
* Estimated pulmonary artery pressure ≥35mmHg
* Hemoglobin concentration ([Hgb]) less than 7 g / dL
* Need for invasive ventilation during preoperative immediate post-extubation defined in the preoperative period
* Patients with obstructive sleep apnea previously treated with CPAP
* Severe psychiatric disorder
* Language barrier

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference in mean PaO2 values after surgery | 24 hours
  Arterial blood samples for blood gas analysis are collected at 1 hour, 2 hours and 24 hours post-extubation. The differences in the mean values of PaO2 are registered and analysed.
Difference in mean PaO2/FiO2 ratio values after surgery | 24 hours
  Arterial blood samples for blood gas analysis are collected at 1 hour, 2 hours and 24 hours post-extubation. The differences in the mean values of PaO2/FiO2 ratio are registered and analysed.

SECONDARY OUTCOMES:
Difference in mean FEV 1 and FVC values | 24 hours
  Spirometry is performed at 1 hour, 2 hours and 24 hours post-extubation. The differences in the mean values of FEV1 and FVC are measured and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Guimarães, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar Porto, Porto, Portugal